CLINICAL TRIAL: NCT04849936
Title: Diagnostische Genauigkeit fäkaler Biomarker im Vergleich Zur Endoskopie Mit Und Ohne Konfokaler Laserendomikroskopie in Der Routineversorgung Zur Bestimmung Der Entzündungsaktivität Bei Patienten Mit Gastrointestinalen Diagnosen
Brief Title: A Diagnostic Accuracy Study Testing Fecal Biomarkers In Comparison To Endoscopic Examination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Sozialstiftung Bamberg (Other); Enterosan Labor LS SE & Co.KG (Unknown)
Responsible Party: Principal Investigator, Jost Langhorst, Prof. Dr. med., Universität Duisburg-Essen
Other Study IDs: 20025
Record Dates: First submitted 2020-10-02; First posted 2021-04-19 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Bowel Diseases
Keywords: inflammatory bowel diseases; fecal biomarkers; calprotectin; lactoferrin; pmn-elastase; human beta-defensin; zonulin
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- evaluation of fecal biomarkers: comparison of the biomarker levels between different gastrointestinal diseases
  Interventions: Diagnostic Test: Testing Fecal Biomarkers In Comparison To Endoscopic Examination With Confocal Laser Endomicroscopy

INTERVENTIONS:
Diagnostic Test: Testing Fecal Biomarkers In Comparison To Endoscopic Examination With Confocal Laser Endomicroscopy — Patients, who were examined during a routine diagnostics, should submit an extra morning stool sample up to two weeks before or after the gastroscopy and/or coloscopy to generate the data of the fecal biomarker mentioned above.

SUMMARY:
In this study it will be explored whether the levels of fecal biomarkers are associated with histologic inflammation of the intestinal mucosa and concomitant alteration of the mucosal permeability. The aim of the study is to assess the diagnostic accuracy of fecal biomarkers especially to detect the potential of differentiation between inflammatory and functional gastrointestinal diseases.

The following biomarkers will be examined in the stool of the participants: calprotectin, lactoferrin, pmn-elastase, human beta-defensin, zonulin, alpha-antitrypsin.

DETAILED DESCRIPTION:
For this study inpatients and outpatients of the clinic for integrative medicine and naturopathy Bamberg, Germany, who had a routine gastroscopy and/or coloscopy with tissue biopsy or an endoscopy with confocal laser endomicroscopy and tissue biopsy were enclosed.

These patients, who were examined during a routine diagnostics, should submit an extra morning stool sample up to two weeks before or after the gastroscopy and/or coloscopy to generate the data of the fecal biomarker mentioned above.

On the basis of the biopsy samples generated through the routine examination we can determine the histology scores, Nancy Index and Riley Score. The determined scores, the data of the fecal biomarkers and the results of the confocal laser endomicroscopy as well as, if available, more clinical data such as the clinical activity index (CAI), the MAYO-Score/Disease Activity Index (DAI), the endoscopic Rachmilewitz-Index (REI) and the Questionnaire for inflammatory bowel disease (IBDQ) will be anonymised inserted into a SPSS data bank and will then be interpreted.

For the adequate description of the collective data of gender, age, blood levels and medication will be gathered and added to the data bank anonymised.

The calculated data will then be compared with the clinical evaluation of the patients with symptomatic irritable bowel syndrome, active inflammatory bowel diseases and patients with other gastrointestinal diseases.

The aim of this study is to develop improved methods for non invasive diagnostics of gastrointestinal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Signed declaration of consent
* Presence of a confirmed diagnosis of

  1. Inflammatory bowel diseases
  2. Irritable bowel syndrome
  3. Gastrointestinal diseases, except participants with diagnosis of group 1 or 2 (e.g. celiac disease, food allergies, microscopic colitis, diverticulosis, diverticulitis)
  4. Healthy controls as part of a preventive medical check-up

Exclusion Criteria:

* No indication for endoscopic examination as part of routine care
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with inflammatory bowel disease, patients with symptomatic non-inflammatory bowel disease, and patients with other gastrointestinal diseases who routinely undergo endoscopic examination at the center in the form of endoscopy with tissue biopsies with and without confocal laser endomicroscopy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
correlation analyses | data of biomarkers generated two weeks before or two weeks after the gastroscopy and/or coloscopy
  Correlation analyses will be performed to determine if there is a correlation between fecal biomarker values and confocal laser endomicroscopy results and histologic scores. If available, correlations between the fecal biomarkers and other parameters such as clinical activity index (CAI), Mayo score/disease activity index (DAI), endoscopic Rachmilewitz index (REI), and inflammatory bowel disease questionnaire (IBDQ) data will also be calculated.
  In addition, group comparisons will be performed to test whether fecal biomarkers differ between (1) the different levels of the Nancy index and (2) the classification into "patients in remission" and "patients with disease activity" given according to histological assessment. Receiver operating characteristic (ROC) curves will also be used to determine optimal cut-offs and calculate sensitivity and specificity of fecal biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Sozialstiftung Bamberg, Klinik für Intergrative Medizin, Bamberg, Bavaria, Germany